CLINICAL TRIAL: NCT03733808
Title: Repetitive Transcranial Magnetic Stimulation (rTMS) of the Dorsolateral Prefrontal Cortex for the Treatment of Gambling Disorder: a Pilot Study
Brief Title: High Frequency rTMS Over l-DLPFC in Gambling Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione Novella Fronda (Other)
Collaborators: Casa di Cura Park Villa Napoleon (Unknown); University of Padova (Other); Istituto Italiano di Tecnologia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: rTM20NG4MBLDSD
Record Dates: First submitted 2018-11-06; First posted 2018-11-07 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Gambling Disorder
Keywords: rTMS
MeSH Terms: conditions — Gambling | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Double blind, randomized, sham-controlled with a 1:1 allocation into 2 parallel arms
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active rTMS treatment (Active Comparator): Active High frequency rTMS will be administered with a Magventure MagPro Stimulator R30 using a butterfly coil. The stimulation protocol parameters will be set as follow: frequency of 15 Hz, of 100% of resting motor threshold (rMT), 40 trains, 60 pulses per train, 15 s intertrain-interval, 2400 pulses per session.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation
- Sham rTMS treatment (Sham Comparator): Sham rTMS will be administered with a Magventure MagPro Stimulator R30 using a butterfly sham coil. The same procedures of active High frequency rTMS will be used.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation — Non-invasive brain stimulation technique

SUMMARY:
Gambling disorder (GD), currently considered a behavioral addiction, show substantial similarities with substance use disorders (SUDs) in terms of neurobiology and symptomatology. In particular, alterations in prefrontal control circuit may underlie vulnerability to gambling- and drug-related cues and diminished cognitive control over craving, and negative emotions. Repetitive transcranial magnetic stimulation (rTMS) of the dorsolateral prefrontal cortex (DLPFC) could represent a novel approach to remodel these brain circuits.

The aim of this study is to evaluate High frequency (HF) rTMS over the left DLPFC as an efficacious treatment for reduction of gambling urges and behavior in a randomized double-blind placebo-controlled design in which 36 GD patients will receive active or sham rTMS for 12 weeks.

DETAILED DESCRIPTION:
Gambling disorder (GD) is a progressive and recurrent maladaptive pattern of gambling behavior, leading to impaired functioning.

GD has been recategorized from an impulse control disorder to an addiction-related disorder in the fifth edition of Diagnostic and Statistical Manual of Mental (DSM-5) reflecting the growing evidence of the substantially overlapping between the neurobiology of GD and substance use disorders (SUDs). Both GD and SUDs are characterized by malfunction in reward, stress and cognitive-control circuits, which underlie manifestations such as compulsive gambling or compulsive drug consumption, craving, altered reward sensitivity, impaired self-control and decision-making processes. Particularly, similar alterations in cortico-limbic-striatal and prefrontal control circuits have been shown associated to the emergence of drug cravings and gambling urges. Hence, craving might be seen as a core component across addictions. Indeed, identifying and targeting the neurocircuit alterations underlying craving, may allow to treat this feature across different addictions with similar strategies.

In this regard, High frequency (HF) repetitive transcranial magnetic stimulation (rTMS) over the left dorsolateral prefrontal cortex (l-DLPFC), is a promising approach for modulating brain circuits underlying cue-induced craving. Since alterations in these circuits have been shown to underlie the emergence of gambling urges, HF rTMS may represent a potential treatment also for GD patients.

Thus, the main goals of this clinical trial are to 1) assess whether HF rTMS over l-DLPFC reduces urges to gamble and problem behaviors gambling related; 2) investigate whether rTMS induces hemodynamics changes in DLPFC activity in response to specific tasks that elicit such areas as visual stimuli associated with gambling; 3) assess whether rTMS induces improvements in decision making processes of GD patients; and 4) evaluate the effects of HF rTMS over l-DLPFC on resting functional connectivity, focusing mainly in connectivity changes of cortical and subcortical regions involved in this disorder.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65;
* Current DSM-5 diagnosis of Gambling Disorder;
* Right-handed;

Exclusion Criteria:

* Current DSM-5 diagnosis of Schizophrenia Spectrum and other Psychotic Disorders;
* Current DSM-5 diagnosis of Bipolar and related Disorders;
* Use in the past 4 weeks of any medication with known pro-convulsant action; or current regular use of any psychotropic medications (benzodiazepines, antipsychotic medications, tricyclic antidepressants, anti-epileptics, mood stabilizers);
* Any history of any clinically significant neurological disorder, including organic brain disease, epilepsy, stroke, brain lesions, multiple sclerosis, previous neurosurgery, or personal history of head trauma that resulted in loss of consciousness for > 5 minutes and retrograde amnesia for > 30 minutes;
* Any personal history of seizures other than febrile childhood seizures;
* Presence of iron magnetic objects in the body contraindicated for treatments with rTMS and for participation in MRI sessions (pacemakers or other electrical devices implants, brain stimulators, some types of dental implants, aneurysm clips, metal implants, permanent eyeliner, fragments of projectile);
* Inability to remain lying on the back for up to 2 hours in the MRI plant;
* Current DSM-5 diagnosis of any Substance Use disorder with the exception of Tobacco Use Disorder and Mild Alcohol Use Disorder;
* Positive drug urine test to one or more classes of substances of abuse;
* For female subjects: pregnancy or breastfeeding in progress;
* Judicial provision that includes a cure in progress or if the subject is already engaged in a cure for gambling disorder;
* Any psychiatric, medical or social condition whether or not listed above, due to which, in the judgment of the PI and after any consults if indicated, participation in the study is not in the best interest of the patient;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2018-12-11 (Actual); Primary Completion 2021-08 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
High frequency rTMS effects on changes of the gambling symptoms severity | Baseline- Day 30 (after 16 rTMS sessions)- Day 60 (after 24 rTMS sessions)- Day 90 (after 32 rTMS sessions)- after 1 month follow-up- after 2 months follow-up- after 3 months follow-up
  The main outcome will be defined as the difference in the variation between baseline and after treatment day 30 of the severity of gambling symptoms assessed through the G-SAS (Gambling Symptom Assessment Scale). Range from: 0-48 (higher values=worse symptoms)

SECONDARY OUTCOMES:
High frequency rTMS effects on prefrontal hemodynamics activity in response to cue reactivity tasks | Baseline- Day 30 (after 16 rTMS sessions)- Day 60 (after 24 rTMS sessions)- Day 90 (after 32 rTMS sessions)- after 1 month follow-up- after 2 months follow-up- after 3 months follow-up
  Functional near-infrared spectroscopy (fNIRS) assessment during cue reactivity task
High frequency rTMS effects on the propensity for future reinforcers to maintain current responding | Baseline- Day 30 (after 16 rTMS sessions)- Day 60 (after 24 rTMS sessions)- Day 90 (after 32 rTMS sessions)- after 1 month follow-up- after 2 months follow-up- after 3 months follow-up
  This decision making process will be evaluated through delay discounting paradigm. Basing on subject's responses and using of a hyperbolic function an k index will be calculate, indicating the rate with which the subjective value declines: smaller values (close to 0) indicate a preference for postponed rewards, larger values (> 0.5) indicate a preference for immediate rewards.
High frequency rTMS effects on changes in decision-making ability linked to emotional and activation self-regulation functions | Baseline- Day 30 (after 16 rTMS sessions)- Day 60 (after 24 rTMS sessions)- Day 90 (after 32 rTMS sessions)- after 1 month follow-up- after 2 months follow-up- after 3 months follow-up
  This decision making process will be evaluated through Iowa Gambling Task. Two types of indices will be calculated that measure participants' a) tendency to choose advantageously (where the choice of decks is likely to yield smaller rewards for each card drawn, but minimizes larger losses, over time) and their b) tendency to select from decks that offer infrequent (though larger) loss.
High frequency rTMS effects on resting functional connectivity | Baseline- Day 90 (after 32 rTMS sessions)
  Functional MRI assessment

CONTACTS AND LOCATIONS:
Overall Officials: Franco Garonna, MD, Principal Investigator — Casa di Cura Park Villa Napoleon; Stefano Cardullo, PhD, Study Chair — Fondazione Novella Fronda
Locations (1):
- Casa di Cura Park Villa Napoleon, Preganziol, Treviso, Italy